CLINICAL TRIAL: NCT01375504
Title: Enhancing Self Regulation With Mindfulness Training and Its Effect on Body Mass Index and Cardiovascular Risk Markers in Obese Adults: A Randomized Pilot Clinical Trial
Brief Title: Effect of Self Regulation With Mindfulness Training on Body Mass Index and Cardiovascular Risk Markers in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amit Sood, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-001775
Record Dates: First submitted 2011-06-13; First posted 2011-06-17 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Obesity
Keywords: Obesity; Body Mass Index; Mindfulness Training; Attention and Interpretation Therapy
MeSH Terms: conditions — Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Counseling (Active Comparator): The control group will receive two sessions of dietary counseling (with instruction to follow a weight loss program) provided by a clinical dietician, consistent with current routine care for adults with obesity.
  Interventions: Behavioral: Dietary Counseling
- Mindfulness Training Program (Other): The mindfulness training program will be administered over three 90-minute sessions by a physician and clinical dietician with expertise in mind-body medicine and nutrition.
  Interventions: Behavioral: Mindfulness Training Program

INTERVENTIONS:
Behavioral: Dietary Counseling — The control group will receive two sessions of dietary counseling (with instruction to follow a weight loss program) provided by a clinical dietician, consistent with current routine care for adults with obesity.
  Arms: Dietary Counseling
Behavioral: Mindfulness Training Program — The mindfulness program will be administered over three 90-minute sessions by a physician and clinical dietician with expertise in mind-body medicine and nutrition.
  Arms: Mindfulness Training Program

SUMMARY:
This study is designed to assess the effect of a mindfulness training program with special focus on diet and nutrition vs. dietary counseling in 40 obese adults (BMI range 30-40) and their partner/spouses (irrespective of their BMI), in a 6-month pilot randomized controlled trial.

DETAILED DESCRIPTION:
Obesity is associated with deficits in self regulation. Approaches that foster increased non-judgmental present moment awareness and increased acceptance have been demonstrated to enhance self regulation. One commonly used approach that synthesizes these concepts is mindfulness training. This study is designed to assess the effect of a mindfulness training program with special focus on diet and nutrition, on body mass index, cardiovascular risk markers, peripheral blood telomere length and telomerase levels in obese adults. The mindfulness training program is adapted from the Attention and Interpretation Therapy developed by study investigators at Mayo Clinic. The study is designed as a 6-month pilot randomized controlled trial involving 40 obese adults and their partners/spouses with standard dietary counseling as the control intervention. Promising feasibility and efficacy data from the study will prompt us to pursue a larger, multi-center trial to more definitively test this program as well as apply this intervention in clinical practice.

ELIGIBILITY:
PRIMARY PARTICIPANT

Inclusion Criteria:

* Obese adults (BMI ≥ 30)
* Currently working at Mayo Clinic Rochester
* Able to provide informed consent
* Stable weight (within + 10 pounds) during the three months prior to enrolling in the study

Exclusion Criteria:

* Currently (in the past six months) attending a weight loss program
* Underlying genetic or endocrine cause for weight gain
* Current cancer
* Medications known to affect weight (corticosteroids, antidepressants, anti psychotics, mood stabilizers, and anti-epileptic medications)
* Musculoskeletal conditions affecting the ability to adequately perform general physical activity
* Active smoking
* Substance abuse
* Quitting smoking within 6 months of enrolling in the study
* Have clinically significant acute unstable neurological, psychiatric, hepatic, renal, cardiovascular or respiratory disease that will prevent participation in the study
* Have an established practice of meditation for three or more months
* Not willing to complete study outcome measures.

PARTNER/SPOUSE

Inclusion Criteria:

* Able to provide informed consent

Exclusion Criteria:

* Have clinically significant acute unstable neurological,Psychiatric, hepatic, renal, cardiovascular or respiratory disease that will prevent participation in the study
* Have an established practice of meditation for three or more months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline to a healthier lifestyle. | 6 Months
  Improvement in general health.

SECONDARY OUTCOMES:
Change from baseline in vital signs. | 6 Months
  Body mass index (BMI) and absolute and percentage weight loss will be compared.
Change from baseline in laboratory values. | 6 Months
  Peripheral blood telomere length and telomerase levels, and cardiovascular risk markers will be compared.
Change from baseline in stress management. | 6 Months
  Stress, anxiety, and quality of life will be measured on various study questionnaires.
Change in baseline on different aspects of eating. | 6 Months
  Mindful eating, self efficacy and self regulation in eating will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sood, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States